CLINICAL TRIAL: NCT04819672
Title: Effect of Low Intensity Resistance Training Combined With Partial Blood Flow Restriction on Pain and Function in Individuals With Knee Osteoarthritis: a Randomized Controlled Study
Brief Title: Effect of Low Intensity Training Combined With Partial Restriction of Blood Flow in Individuals With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, PhD, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PIBIC_Riccelli
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Ischemic Preconditioning; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity Training associated with Partial Blood Flow (Experimental): In the experimental group, a cuff with compression at 60% of the pressure required for total arterial occlusion will be placed, 16 treatment sessions in 8 weeks: warm-up, stretching of the lower limbs, strengthening of the quadriceps (knee extension and squat). The cuff with partial blood flow restriction will be used during knee extension and squat exercises.
  Interventions: Other: Low Intensity Training associated with Partial Blood Flow
- Low Intensity Training associated with Partial Blood Flow-Sham (Sham Comparator): In the sham group, the cuff will be placed, but there will be no arterial occlusion pressure, 16 treatment sessions in 8 weeks: warm-up, stretching of the lower limbs, strengthening of the quadriceps (knee extension and squat). The cuff without partial blood flow restriction will be used during knee extension and squat exercises.
  Interventions: Other: Low Intensity Training associated with Partial Blood Flow-Sham

INTERVENTIONS:
Other: Low Intensity Training associated with Partial Blood Flow — 16 treatment sessions in 8 weeks: warm-up, stretching of the lower limbs, strengthening of the quadriceps, hamstrings, sural triceps, abductors and adductors of the hip. The Partial blood flow restriction will be used during knee extension and squat exercises. During the exercises, a metronome will be used for the time under tension, 2 seconds for the eccentric and concentric phase.
  Arms: Low Intensity Training associated with Partial Blood Flow
Other: Low Intensity Training associated with Partial Blood Flow-Sham — 16 treatment sessions in 8 weeks: warm-up, stretching of the lower limbs, strengthening of the quadriceps, hamstrings, sural triceps, abductors and adductors of the hip. The Partial blood flow restriction will be used during knee extension and squat exercises. During the exercises, a metronome will be used for the time under tension, 2 seconds for the eccentric and concentric phase.
  Arms: Low Intensity Training associated with Partial Blood Flow-Sham

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative infection that presents clinical features such as pain and limited range of motion. A weakness of the quadriceps makes this joint more susceptible to wear and tear to the articular cartilage, especially in the medial compartment of the knee. As a result, it is necessary to promote an increase of at least 30% in quadriceps strength for a beneficial effect on pain and 40% in functional capacity. Therapeutic exercises are used to increase strength muscle, in addition to high intensity exercises, to decrease joint pain, low to moderate intensity resistance training has been included, with the new approach of using partial blood flow restriction.

DETAILED DESCRIPTION:
Physical therapy sessions will be individual and supervised, will last 30-40 minutes, twice a week, for eight weeks.

Participants will warm up with a walk or bike for 5 minutes. Then, a single series of sustained stretching will be performed for a period of 40 seconds for the following muscle groups: hamstrings, quadriceps femoris, hip abductors, hip adductors and gastrocnemius. After the stretches, active muscle strengthening exercises will be performed focusing on the quadriceps femoris muscle. The knee extension and squat exercises will be performed in four sets, with the first set being thirty repetitions or even volitional fatigue, and the following three sets will be fifteen to twenty-four repetitions, with 90 seconds of rest between each series, and two minutes of rest at the end of the four series. Both groups will perform these exercises with 30% of 1RM. The maximum load that will be lifted until volitional fatigue between 7 to 10 repetitions will be used instead of direct 1RM measurement.

Regarding the intensity of the exercises, this will be monitored by the physical therapist according to the perception of the level of effort and difficulty reported by the participant when completing the series of knee extension and squat, according to the specifications of the modified Borg scale (CR-10) . The exercises will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant. The load will be increased by 2-10% when the patient is able to perform 24 complete repetitions in the last series of the exercise with perceived effort <60%. During the exercises, a metronome will be used for the time under tension, 2 seconds for the eccentric and concentric phase.

Partial blood flow restriction will be used during knee extension and squat exercises as follows: Arterial occlusion pressure will be measured by placing a cuff on the proximal thigh in a standing position. The measurement of insufflation for each patient will be established as follows: with the participant in the supine position, the pulse of the pedal will be located with the LOGIQ e (GE Healthcare) Ultrasound. The cuff pressure will be increased until the pedal pulse can no longer be identified, and then the arterial occlusion pressure will be recorded when the pulse is restored. The RPFS will be performed at 60% of the arterial occlusion pressure for the experimental group and there will be no arterial occlusion pressure for the sham group.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of clinical diagnosis of osteoarthritis according to the criteria established by the American College of Rheumatology;
* OA knee radiograph grades 2 - 4 according to the Kellgren-Lawrence scale;
* Reporting knee pain with minimum intensity of 3 on Numerical Pain Scale;
* Complaints of pain and functional reduction in the last three months;

Exclusion Criteria:

* Diabetes type I or decompensated;
* Peripheral vascular disease;
* Uncontrolled hypertension;
* History of deep vein thrombosis;
* History of stroke;
* History of cancer;
* Cardiac pacemaker;
* Cognitive disorders;
* Neurological deficits (sensory or motor)
* Body mass index above 40 kg/m2
* Hip symptomatic osteoarthritis
* Low back pain
* Use of painkillers in the last 24 hours;
* Intra-articular infiltration with hyaluronic acid and corticosteroids in the last 6 months;
* Orthopedic surgery on lower limbs;
* Systemic inflammatory disease;
* Not able to walk

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain subscale - Knee Injury and Osteoarthritis Outcome Score | 8-week follow-up
  Pain subscale - KOOS was assessed, where 0 corresponded to no pain and 100 corresponded to worst pain.
Activities of daily living subscale - Knee Injury and Osteoarthritis Outcome Score | 8-week follow-up
  Activities of daily living subscale - KOOS was assessed, where 0 corresponded to normal function and 100 corresponded to worst function.
Numeric Pain Scale | 8-week follow-up
  Pain was assessed by use of an 11-point Numeric Pain Scale, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain.

SECONDARY OUTCOMES:
Timed Up And Go Test (TUG-Test) | 4- and 8-weeks follow-up
  This test quantifies the functional capacity in seconds by the time the individual needs to perform the task of getting up from a chair with a backrest without the aid of arms, walking three meters, turning, going back to the chair and sitting again, wearing regular shoes and without walking assist devices. A tape will be used to mark the distance of three meters. The patient will perform a practical test and two effective tests, assuming the shortest time for statistical analysis.
30 Seconds Chair Stand Test | 4- and 8- weeks follow-up
  This test quantifies the maximum number of repetitions that the individual is able to get up and sit without using the armrest in a 44 cm chair in a period of 30 seconds. The patient must have his arms crossed over his chest and his feet at the shoulder line to perform the test.
Global Perceived Effect Scale | 4- and 8- weeks follow-up; and 6-month follow up
  Scale of 11 points ranging from minus five points (extremely worse), zero (no change) to five points (completely recovered). For all measures of the perceived global effect, participants will be asked: "compared to starting treatment, how would you describe your knee today?". Positive scores represent better recovery, negative scores indicate worsening of symptoms and zero without change.
Assessment of strength of the quadriceps femoris using the isokinetic dynamometer | 4- and 8-weeks follow-up
  Strength assessment will be measured by the Isokinetic Dynamometer by a blind assessor. The positioning will be carried out as follows: when seated in the chair, the popliteal fossa will be positioned 2 cm from the end of the seat, the hip positioned at 85 ° of flexion, the axis of movement of the device was aligned with the intercondylar line of the knee, and the lever arm kept 2 cm above the lateral malleolus. Belts will be placed to stabilize the trunk, abdomen and thigh of the evaluated member. After that, the limits of maximum range of motion and flexion will be established, the adequacy of the initial knee position at 90° of flexion and the weighing of the lower limb to be evaluated. The participant will be registered in the device system, with information such as dominance and limb injury. The protocol that will be used involves five concentric repetitions with maximum intensity at 60 °/s for strength assessment.
Numeric Pain Scale | 4-week and 6-month follow-up
  Pain was assessed by use of an 11-point Numeric Pain Scale, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain
Pain subscale - Knee Injury and Osteoarthritis Outcome Score | 4-week and 6-month follow-up
  Pain subscale - KOOS was assessed, where 0 corresponded to no pain and 100 corresponded to worst pain.
Activities of daily living subscale - Knee Injury and Osteoarthritis Outcome Score | 4-week and 6-month follow-up
  Activities of daily living subscale - KOOS was assessed, where 0 corresponded to normal function and 100 corresponded to worst function.
Others subscales - Knee Injury and Osteoarthritis Outcome Score | 4- and 8-weeks follow-up; and 6-month follow up
  It contains 42 items, divided into five subscales: other symptoms (7 questions), function in sport (5 questions) and recreation and quality of life related to the knee (4 questions) ). Its score ranges from 0 (extreme problem) to 100 (without problems) separately within each subscale.
Amount of non-hormonal anti-inflammatory and/or analgesics ingested | 4- and 8-weeks follow-up; and 6-month follow up
  The amount of non-hormonal anti-inflammatory drugs and/or painkillers will be counted as clinical outcomes in all assessments.